CLINICAL TRIAL: NCT01246882
Title: Stroke Inpatient Rehabilitation Reinforcement of ACTivty: An International Multisite Clinical Trial
Brief Title: Stroke Inpatient Rehabilitation Reinforcement of ACTivity
Acronym: SIRRACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Taiwan University Hospital (Other); Washington University School of Medicine (Other); University of Vigo (Other); Morinomiya Hospital, Osaka, Japan (Unknown); Mayo Clinic (Other); IRCCS San Camillo, Venezia, Italy (Other); Fairlawn Hospital, Worcester, MA, USA (Unknown); Chonnam National University Hospital (Other); Ain Shams University (Other); MedStar National Rehabilitation Network (Other); St. Luke's Hospital, Pennsylvania (Other); Father Muller Medical College (Other); Burke Rehabilitation Hospital (Other); Burwood Hospital, Christchurch, New Zealand (Other); Gazi University (Other); University College Hospital, Ibadan, Nigeria (Unknown); Rehabilitation Hospital, Barcelona, Spain (Unknown); IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bruce H. Dobkin, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-000134
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: Stroke, gait, walking, disability; wireless inertial sensing; mobile health
MeSH Terms: conditions — Stroke | interventions — Accelerometry; Telemedicine; Physical Therapy Modalities; Stroke Rehabilitation; Locomotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Augmented activity feedback (Experimental): Feedback three times per week about 10-m walking speed, plus amount and types of physical activity measured using wireless bilateral ankle sensors that detect bouts of walking and cycling speed, duration, and distance.
  Interventions: Behavioral: Augmented activity feedback
- speed-only feedback (Active Comparator): Feedback three times per week about overground walking speed over 10 meters.
  Interventions: Behavioral: Speed-only feedback

INTERVENTIONS:
Behavioral: Augmented activity feedback — Feedback about walking speed and amount of physical activity will be provided 3 times per week from data acquired from wireless sensors on each ankle.
  Other Names: accelerometry; hemiparetic stroke; mobile health; wireless health; feedback about performance; physical therapy for stroke rehabilitation; locomotion
  Arms: Augmented activity feedback
Behavioral: Speed-only feedback — Feedback about walking speed will be provided 3 times per week.
  Arms: speed-only feedback

SUMMARY:
The purpose of this study is to determine the effects of daily feedback about physical activity (number of bouts of walking, duration of bouts, total walking distance, average and fastest walking speed) and walking average speed compared to feedback about walking speed only on walking-related outcomes during inpatient rehabilitation for stroke. For the first time, daily walking and other exercise will be monitored by bilateral triaxial accelerometers on the ankles. Activity-recognition algorithms will analyze the inpatient sensor data and return a summary to the participants at each site.

DETAILED DESCRIPTION:
Wireless Sensor System The inertial sensor system and activity-recognition algorithms were previously described and tested for short-term reliability. Three sets of triaxial accelerometers (Gulf Coast Data Concepts, Waveland, MS) were mailed to each site's coordinator. Therapists placed one sensor on each ankle before participants got out of bed each morning and removed them once they were in bed at the end of the day; sensor use during weekends was optional. A soft snap band secured each sensor proximal to the medial malleolus, flush against the bony tibia. Every night, sensors were plugged into a local computer to recharge while accelerometer data were uploaded to the central server at UCLA for secure storage and processing. Sensor Calibration and Data Processing In recognition of the variations in gait speed and stand and swing symmetry that occur in patients who need inpatient rehabilitation after stroke, we chose to generate individual templates of each participant's gait from a pair of standardized walks. On study entry participants performed two stopwatch- timed 10-meter walks at self-selected casual and safest fast walking speeds. A hybrid classifier employing dynamic time warping and Naïve Bayes algorithms generated statistical models of each participant's gait based on the two walks. Repeat walks were performed and the templates updated weekly for the remainder of each participant's rehabilitation stay to account for expected changes in gait parameters.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute inpatient rehabilitation of a first stroke (or second stroke after full recovery from prior TIA/Stroke)
* Time from onset of stroke to admission for rehabilitation < 35 days
* Stroke from any cause (thrombotic infarct, cardioembolus, intracerebral hemorrhage) that includes unilateral hemiparesis. Hemiparesis means less than / equal to 4/5 strength by the British Medical Council scale for hip flexion tested supine and for knee or ankle flexion and extension (scores less than / equal to 22 of 25 possible points)
* Ability to follow simple instructions, especially to understand verbal reinforcement about activity.
* Independent in mobility prior to admission by the Barthel Index.
* Able to walk with no more than physical assistance of 2 persons for at least 5 steps (for example, 3 strides of the left leg alternating with 2 on the right leg). Subjects can use any type of assistive device and brace needed.
* Able to understand and repeat information related to the Informed Consent. The subject signs a Consent form.

Exclusion Criteria:

* Current medical disease that will limit physical therapy at the time of randomization or limited walking prior to the stroke, such as serious infection, DVT, orthostatic hypotension, > stage 2 decubitus ulcer of buttocks or legs, congestive heart failure, claudication, and pain with weight-bearing or walking. Subjects can be entered if a complication resolves within 7 days of admission screening.
* Aphasia with inability to follow 2-step directions during therapeutic instructions or answers Yes/No to questions with < 75% accuracy related to personal health and symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Gait speed | Discharge

SECONDARY OUTCOMES:
Distance walked in 3 minutes | Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H Dobkin, MD, Principal Investigator — University of California, Los Angeles
Locations (18):
- United States (5):
  - Fairlawn Hospital, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Burke Rehabilitation Hospital, White Plains, New York
  - St. Luke's Hospital, Allentown, Pennsylvania
- Ain Shams University, Cairo, Egypt
- Father Muller Medical College, Karnataka, India
- National Rehabilitation Hospital, Dublin, Ireland
- Italy (2):
  - San Raffaele Hospital, Milan
  - Sam Camillo, Venice
- Morinomiya Hospital, Osaka, Japan
- Burwood Hospital, Christchurch, New Zealand
- Univeristy College Hospital, Ibadan, Nigeria
- Chonnam National Hospital, Gwangju, South Korea
- Spain (2):
  - Rehabilitation Hospital, Barcelona
  - University of Vigo, Vigo
- National Taiwan University Hospital, Taipei, Taiwan
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Dobkin BH, Dorsch A. The promise of mHealth: daily activity monitoring and outcome assessments by wearable sensors. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):788-98. doi: 10.1177/1545968311425908. PMID 21989632
- [Result] Dorsch AK, Thomas S, Xu X, Kaiser W, Dobkin BH; SIRRACT investigators. SIRRACT: An International Randomized Clinical Trial of Activity Feedback During Inpatient Stroke Rehabilitation Enabled by Wireless Sensing. Neurorehabil Neural Repair. 2015 Jun;29(5):407-15. doi: 10.1177/1545968314550369. Epub 2014 Sep 26. PMID 25261154